CLINICAL TRIAL: NCT04303065
Title: Dexamethasone for the Treatment of Traumatic Brain Injured Patients With Brain Contusions and Pericontusional Edema: Study Protocol for a Prospective, Randomized and Double Blind Trial.
Brief Title: Trial of Dexamethasone for Traumatic Brain Injured Patients With Brain Contusions and Pericontusional Edema
Acronym: DEXCON-TBI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped because of lack of funding
Sponsor: Jon Pérez Bárcena (Other)
Collaborators: Fundación Mutua Madrileña (Other); Sociedad Española de Medicina Intensiva, Crítica y Unidades Coronarias (SEMICYUC) (Unknown)
Responsible Party: Sponsor-Investigator, Jon Pérez Bárcena, MD, Hospital Son Espases
Organization: Hospital Son Espases (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-004038-41
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Brain Injury; Cerebral Edema; Head Injury Trauma
Keywords: traumatic; brain; injury; contusion; edema; steroids
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema; Wounds and Injuries; Contusions; Edema | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the pharmacist, who masks the capsules and labels the containers, will know the assignement of the codes, and will keep them blind until the last phase of the study, after the main statistical analysis, or when unmasking is required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone will be a short and descending course: 4mg/6 hours (2 days); 4 mg/8 hours (2 days); 2 mg/6 hours (2 days); 2 mg/8 hours (2 days); 1 mg/8 hours (2 days); 1 mg/12 hours (2 days).
  Dexamethasone (Fortecortin®) will be acquired from ERN, SA. Laboratories (Barcelona, Spain). The Son Espases Pharmacy Department will be in charge of developing and conditioning the 4mg, 2mg and 1mg dexamethasone / placebo capsules needed for 12 days of treatment, keeping the researchers blind
  Interventions: Drug: Dexamethasone Oral
- Control (Placebo Comparator): The preparation and conditioning of the capsules will be carried out following the standardized work procedures of the pharmaceutical laboratory and its quality controls, previously authorized by the Agencia Española del Medicamento (AEMPS).
  The Son Espases Pharmacy Department will be responsible for identifying the containers and sending them by courier to the participating hospitals. A record of the dispensing of test samples will be kept and will be sent in acknowledgment of receipt for control
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Dexamethasone Oral — It will be a short and descending course of oral dexamethasone: 4mg/6 hours (2 days); 4 mg/8 hours (2 days); 2 mg/6 hours (2 days); 2 mg/8 hours (2 days); 1 mg/8 hours (2 days); 1 mg/12 hours (2 days).
  Arms: Dexamethasone
Drug: Placebo oral tablet — The preparation and conditioning of the placebo capsules will be carried out following the standardized work procedures of the pharmaceutical laboratory and its quality controls, previously authorized by the Agencia Española del Medicamento (AEMPS).
  Arms: Control

SUMMARY:
The DEXCON-TBI trial is a multicenter, pragmatic, randomized, triple-blind, placebo controlled trial to quantify the effects of the administration of dexamethasone on the prognosis of TBI patients with brain contusions and pericontusional edema. Adult patients who fulfil the elegibility criteria will be randomized to receive dexamethasone or placebo. Patients who have suffered a head injury and have one or more cerebral contusions with visible pericontusional edema in the CT scan can be included in the study. The doses of dexamethasone will be a short and descending course: 4mg/6 hours (2 days); 4 mg/8 hours (2 days); 2 mg/6 hours (2 days); 2 mg/8 hours (2 days); 1 mg/8 hours (2 days); 1 mg/12 hours (2 days). The primary outcome is the Glasgow Scale Outcome Extended (GOSE) performed one month and 6 months after trauma. Other secondary outcomes are: compare the number of episodes of neurological deterioration; compare the symptoms associated with TBI; compare the presence of adverse events during treatment; compare the volume of pericontusional edema before and after 12 days of treatment in both groups of patients; and compare the results of the neuropsychological tests between the two groups of patients one month and 6 months after the TBI. The main analysis will be on an ''intention-to-treat´´ basis. A descriptive analysis of the baseline variables will be made for each treatment group. Logistic regression will be used to estimate the effect of dexamethasone and placebo on GOSE at one month and at 6 months, dichotomized in unfavorable outcome (GOSE 1-6) and favorable outcome (GOSE 7-8). Since the severity of the initial injury will determine significantly the final outcome of the patient, to assess the effect of dexamethasone, efficacy will also be analyzed using the 'sliding dichotomy'. A subgroup analysis will be carried out by stratifying the patients as they present more or less than 10mL of pericontusional edema in the preinclusion CT. We will perform an interim analysis with the patients included during the first year to calculate the conditional power. An independent statistician will blindly perform this analysis. At the same time a safety analysis will be also perfomed. A study with 600 patients would have about 80% power (two sided alpha=5%) to detect a 12% absolute increased (from 50% to 62%) in good outcome.

ELIGIBILITY:
Inclusion Criteria:

* -Patients who have suffered a head injury and have one or more cerebral contusions with visible pericontusional edema in the CT scan.
* Patients with brain contusions in whom non-sugical treatment has been selected initially.
* Age 18 or over and under 85
* Signing of informed consent by the patient or by his legal representative. The fundamental eligibility criterion is the responsible clinician's 'uncertainty' as to whether or not to use dexamethasone in a particular patient with TBI. This pragmatic approach will allow us to see whether the intervention improves patient outcomes under real-life conditions.

Exclusion Criteria:

* Patients with TBI and brain contusions who have required surgery to evacuate the cerebral contusion before randomization.
* Patients with TBI who have required a craniotomy before randomization for any other reason: evacuation of subdural, epidural hematoma or depressed skull fracture.
* Patients with an extracranial Injury Severity Score greater than 18 points.
* Patients in whom the use of corticosteroids is contraindicated.
* Patients who take oral corticosteroids chronically.
* Patients included in another clinical trial.
* Known intolerance or hypersensitivity to dexamethasone.
* Patients with allergy or intolerance to the following excipients contained in dexamethasone / placebo capsules: lactose, corn starch or microcrystalline cellulose.
* Patients with a history of psychotic disorders.
* Patients with inability to take medication orally due to swallowing problems in which it is not indicated to place a nasogastric tube.
* Pregnant or breastfeeding patients.
* Patients in a GCS 3 points situation with bilateral dilated pupils.
* Patients with associated spinal cord injuries.
* Patient with any systemic condition that contraindicates the use of corticosteroids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Glasgow Scale Outcome Extended (GOSE). | one month

SECONDARY OUTCOMES:
Number of episodes of neurological deterioration in both groups of patients during the 12 days of treatment. | 14 days
Symptoms associated with TBI in both groups of patients during the 12 days of treatment. | 14 days
Volume of pericontusional edema before and after 12 days of treatment in both groups of patients. | 14 days
Presence of adverse events between the two groups during the 12 days of treatment. | 14 days
Neuropsychological tests between the two groups of patients one month and 6 months after the TBI. | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moll A, Lara M, Pomar J, Orozco M, Frontera G, Llompart-Pou JA, Moratinos L, Gonzalez V, Ibanez J, Perez-Barcena J. Effects of dexamethasone in traumatic brain injury patients with pericontusional vasogenic edema: A prospective-observational DTI-MRI study. Medicine (Baltimore). 2020 Oct 23;99(43):e22879. doi: 10.1097/MD.0000000000022879. PMID 33120830
- [Background] Lara M, Moll A, Mas A, Picado MJ, Gassent C, Pomar J, Llompart-Pou JA, Brell M, Ibanez J, Perez-Barcena J. Use of diffusion tensor imaging to assess the vasogenic edema in traumatic pericontusional tissue. Neurocirugia (Engl Ed). 2020 Jul 21:S1130-1473(20)30080-4. doi: 10.1016/j.neucir.2020.05.002. Online ahead of print. English, Spanish. PMID 32709492
- [Result] Perez-Barcena J, Castano-Leon AM, Lagares Gomez-Abascal A, Barea-Mendoza JA, Navarro Main B, Pomar Pons J, Perianez Parraga LDM, Ibanez Dominguez J, Chico-Fernandez M, Llompart-Pou JA, Frontera Juan G; DEXCON TBI trial collaborators. Dexamethasone for the treatment of traumatic brain injured patients with brain contusions and pericontusional edema: Study protocol for a prospective, randomized and double blind trial. Medicine (Baltimore). 2021 Jan 22;100(3):e24206. doi: 10.1097/MD.0000000000024206. PMID 33546038

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT04303065/Prot_SAP_000.pdf
  • Study Protocol: Protocol synopsis (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT04303065/Prot_001.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT04303065/Prot_SAP_002.pdf